CLINICAL TRIAL: NCT04292418
Title: Predictors of Rejection in Pediatric Kidney Transplantation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Khalifa, Principle investigator, Assiut University
Other Study IDs: PKTX
Record Dates: First submitted 2020-02-29; First posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Rejection Acute Renal
MeSH Terms: interventions — Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group 1: (rejector group )include Paediatric living donor kidney transplant recipients (aged 4-18 years) at least 35 child recieving standard triple drug immunosuppression consisting tacrolimus an antiproliferative drug [mycophenolate mofetil (MMF) and steroids, with biopsy proven acute rejection in the study group 1 measuring tacrolimus level by elisa test then correlated with hematocrit level measuring mycophenolic acid by elisa test
  Interventions: Drug: Tacrolimus capsule , mycophenolic acid
- study group 2: the second group (non rejector group ) include Paediatric living donor kidney transplant recipients (aged 4-18 years) recieving standard triple drug immunosuppression consisting tacrolimus an antiproliferative drug [mycophenolate mofetil (MMF) and steroids, with biopsy proven acute rejection in the studied group at least 35 child measuring tacrolimus level by elisa test then correlated with hematocrit level measuring mycophenolic acid by elisa test in the study group 2
  Interventions: Drug: Tacrolimus capsule , mycophenolic acid

INTERVENTIONS:
Drug: Tacrolimus capsule , mycophenolic acid — measuring tacrolimus level by elisa test then correlated with hematocrit level measuring mycophenolic acid by elisa test for study group 1 and study group 2

SUMMARY:
Renal transplantation is the best option among the end-stage renal disease (ESRD) treatment alternatives, It is also relatively less expensive than dialysis. Allograft rejection is a major issue in kidney transplantation. Rejection is classified as acute or chronic, cellular or antibody-mediated.Children with kidney transplants require life-long immunosuppressive therapy to prevent rejection of the allograft

DETAILED DESCRIPTION:
The most common medication regimen in the United States includes the combination of corticosteroid (eg, prednisone), a calcineurin inhibitor (or CNI, most commonly tacrolimus), and an antimetabolite such as mycophenolate mofetil (MMF). Cyclosporine and azathioprine are less commonly used for maintenance immunosuppression Tacrolimus level is a main maintenance immunosuppressant in kidney transplantation .In the early days of posttransplant period, hematocrit concentrations are generally low and increase significantly as patient recovers. Because tacrolimus binds strongly to erythrocytes in systemic circulation, the effect of hematocrit on distribution of tacrolimus is important for the methods used to measure tacrolimus concentrations ,hematocrit correction could be a step towards improvement of tacrolimus dose individualization Thearputic drug monitoring of MPA has been proposed to optimize drug dosage avoiding potential hematologic and digestive side effects .MPA monitoring is generally based on the determination of the plasma MPA trough concentration (C0) .

ELIGIBILITY:
Inclusion Criteria:

1. Paediatric living donor kidney transplant recipients (aged 1-18 years)
2. patients received standard triple drug immunosuppression consisting tacrolimus an antiproliferative drug [mycophenolate mofetil (MMF) and steroids
3. recipients with biopsy proven acute rejection in the studied group.

Exclusion Criteria:

1. patients on cyclosporine
2. patients with active infection and dehydration
3. Patients who received multiorgan transplantation Non cooperative patient will be excluded

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Paediatric living donor kidney transplant recipients (aged 1-18 years)
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
predictors of rejection | 2 year
  detect the potentially predictors of rejection in pediatric kidney transplant recipient

SECONDARY OUTCOMES:
measure corrected tacrolimus level and mycophenolic acid | 2 year
  detect the role of corrected tacrolimus level in dose adjustment for better control of immunosuppressive therapy detect the role of neutrophil to lymphocytic ratio in prediction of kidney rejection Role of mycophenolic acid monitoring in prevention of rejection

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bulut IK, Taner S, Keskinoglu A, Sezer TO, Kabasakal C. Pediatric Kidney Transplantation in Patients With Urologic Anomalies. Transplant Proc. 2019 Sep;51(7):2257-2261. doi: 10.1016/j.transproceed.2019.01.155. Epub 2019 Aug 7. PMID 31400969
- [Result] Tamain M, Sayegh J, Lionet A, Grimbert P, Philipponnet C, Hazzan M, Augusto JF, Buchler M, Merlin E, Kosmadakis G, Tiple A, Pereira B, Garrouste C, Heng AE. Extracorporeal photopheresis for the treatment of graft rejection in 33 adult kidney transplant recipients. Transfus Apher Sci. 2019 Aug;58(4):515-524. doi: 10.1016/j.transci.2019.06.031. Epub 2019 Jul 22. PMID 31383541
- [Result] Park WY, Paek JH, Jin K, Park SB, Han S. Long-term Clinical Significance of Tacrolimus Trough Level at the Early Period After Kidney Transplantation. Transplant Proc. 2019 Oct;51(8):2643-2647. doi: 10.1016/j.transproceed.2019.03.065. Epub 2019 Aug 30. PMID 31477420
- [Result] Akbas SH, Ozdem S, Caglar S, Tuncer M, Gurkan A, Yucetin L, Senol Y, Demirbas A, Gultekin M, Ersoy FF, Akaydin M. Effects of some hematological parameters on whole blood tacrolimus concentration measured by two immunoassay-based analytical methods. Clin Biochem. 2005 Jun;38(6):552-7. doi: 10.1016/j.clinbiochem.2005.02.011. PMID 15885236
- [Result] Krischock LA, van Stralen KJ, Verrina E, Tizard EJ, Bonthuis M, Reusz G, Hussain FK, Jankauskiene A, Novljan G, Spasojevic-Dimitrijeva B, Podracka L, Zaller V, Jager KJ, Schaefer F; ESPN/ERA-EDTA Registry. Anemia in children following renal transplantation-results from the ESPN/ERA-EDTA Registry. Pediatr Nephrol. 2016 Feb;31(2):325-33. doi: 10.1007/s00467-015-3201-8. Epub 2015 Sep 18. PMID 26385862
- [Result] Chinnakotla S, Verghese P, Chavers B, Rheault MN, Kirchner V, Dunn T, Kashtan C, Nevins T, Mauer M, Pruett T; MNUM Pediatric Transplant Program. Outcomes and Risk Factors for Graft Loss: Lessons Learned from 1,056 Pediatric Kidney Transplants at the University of Minnesota. J Am Coll Surg. 2017 Apr;224(4):473-486. doi: 10.1016/j.jamcollsurg.2016.12.027. Epub 2017 Feb 27. PMID 28254584
- [Result] Schijvens AM, van Hesteren FHS, Cornelissen EAM, Bootsma-Robroeks CMHHT, Bruggemann RJM, Burger DM, de Wildt SN, Schreuder MF, Ter Heine R. The potential impact of hematocrit correction on evaluation of tacrolimus target exposure in pediatric kidney transplant patients. Pediatr Nephrol. 2019 Mar;34(3):507-515. doi: 10.1007/s00467-018-4117-x. Epub 2018 Oct 30. PMID 30374607
- [Result] Limsrichamrern S, Chanapul C, Mahawithitwong P, Sirivatanauksorn Y, Kositamongkol P, Asavakarn S, Tovikkai C, Dumronggittigule W. Correlation of Hematocrit and Tacrolimus Level in Liver Transplant Recipients. Transplant Proc. 2016 May;48(4):1176-8. doi: 10.1016/j.transproceed.2015.12.096. PMID 27320581